CLINICAL TRIAL: NCT00199927
Title: A Prospective, Randomized, Multicenter Trial Testing the Antiproteinuric Effect of Statins Added to Combined ACE-inhibitor and Angiotensin Receptor Antagonist Therapy in Proteinuric, Chronic Nephropathies
Brief Title: Statins in Proteinuric Nephropathies
Acronym: ESPLANADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Piero Ruggenenti, Mario Negri Institute for Pharmacological Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPLANADE
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Nephropathy; Proteinuria; Hypertension
MeSH Terms: conditions — Proteinuria; Hypertension | interventions — Fluvastatin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard therapy (Active Comparator): Standard therapy
  Interventions: Drug: standard therapy
- fluvastatin (Active Comparator): 40-80 mg/day
  Interventions: Drug: Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin — Starting dose of Fluvastatin of 40 mg/day uptitrated to 80 mg/day
  Arms: fluvastatin
Drug: standard therapy — standard therapy
  Arms: standard therapy

SUMMARY:
End stage renal disease (ESRD) is rapidly growing worldwide. Patients with ESRD have increased morbidity and mortality mostly because of a dramatic excess of cardiovascular disease. Thus, preventing or limiting the progression of chronic nephropathies, in addition to limit the incidence of ESRD, may also postpone death. Drugs that inhibit the renin angiotensin system, such as Angiotensin-Converting-Enzyme inhibitors (ACEi) and Angiotensin II receptor antagonists (ATA), are reno- and cardio-protective in the long-term. There are data that statins,in addition to limit cardiovascular events may have specific reno-protective properties.

Thus we designed a study aimed to evaluate whether statins associated to ACEi and ATA may have an additional reno-protective effect.

ESPLANADE is a multicenter, prospective, randomized, parallel group study in which, after 2 months treatment with ACEi and ATA, two groups of 90 patients, with or without type 2 diabetes, are randomized to 6 months Fluvastatin (40 or 80 mg/day) treatment YES or NO.Twenty Italian Nephrology Units are involved in the trial. The study is fully coordinated by the Clinical Research Center for Rare Disease Aldo e Cele Daccò, Villa Camozzi, Ranica.

DETAILED DESCRIPTION:
INTRODUCTION End stage renal disease (ESRD) is rapidly growing worldwide and costs of providing ESRD care will soon outstrip the available resources. In addition to a poor quality of life, patients with ESRD have 10 to 20 timer higher mortality than age-, race- and gender-matched healthy controls, with > 50% of this excess burden being attributable to cardiovascular risk. Thus, preventing or limiting progression of chronic nephropathies, may serve to limit the incidence not only of ESRD, but also the excess of cardiovascular complications associated with chronic renal disease.

Several data are available that proteinuria is an important determinant of progression to ESRD and a risk factor for increased cardiovascular morbidity and mortality. Drugs, such as Angiotensin-Converting-Enzyme inhibitors (ACEi) and Angiotensin II receptor antagonists (ATA), that decrease proteinuria are also reno- and cardio-protective in the long-term.The combination of these drugs may reduce proteinuria more effectively than the two drugs alone. Preliminary data are also available that statins, in addition to ameliorate the lipid profile may have specific renoprotective properties and, combined to ACEi and ATA, may synergize their antiproteinuric effects in experimental models of chronic renal disease.Moreover, the addition of statins to antihypertensive treatment with or without inhibitors of the renin-angiotensin system has an additive effect on reducing proteinuria also in humans.Whether also in humans combining statins to ACEi and ATA may reduce proteinuria more effectively than ACEi and ATA alone is therefore worth investigating.

AIMS Primary

- To assess whether statins combined to ACEi and ATA more effectively than ACEi and ATA alone reduce urinary protein excretion rate in chronic proteinuric nephropathies.

Secondary

* To assess the effect of statins combined to ACEi and ATA vs. the combination of ACEi and ATA alone on other outcome variables including urinary protein/creatinine ratio, glomerular filtration rate (GFR), lipid profile and, in a subgroup endothelial function. - To evaluate by correlation and multivariate analyses the relationship between baseline /follow-up covariates and the above outcome variables in the study group as a whole and within each treatment group.
* To assess treatment tolerability DESIGN This is be a prospective, randomized, parallel group study in which, following a 2 month Wash-out period from previous treatment (if any) with ACEi, ATA, potassium sparing diuretics or statins, patients will enter a two-month Run-In phase on renin angiotensin system (RAS) inhibitor therapy (ACE inhibition by benazepril for one month and ACE inhibition plus angiotensin II antagonism by combined treatment with benazepril and valsartan for one further month). At completion of the Run-in period and after a baseline evaluation, patients will be randomized to a six-month Treatment period with or without fluvastatin. Regardless of the randomization group, all patients will be offered optimal conservative treatment including optimal blood pressure control(systolic/diastolic blood pressure <130/80 mmHg) and life-style recommendations such as stop smoking and controlled protein and sodium intake.

  180 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* age >16 years
* hypertension, defined as a systolic or diastolic blood pressure > 140 or 90 mmHg respectively (or less in patients with concomitant antihypertensive therapy)
* creatinine clearance >20 ml/min/1.73m2 (with variation of less than 30% in the 3 months prior to study entry)
* urinary protein excretion rate persistently > 1 g/24 hours (average of at least two measurements in two urine collections two weeks apart) without evidence of urinary tract infection or overt heart failure (New York Heart Association class III or more)
* written informed consent

Exclusion criteria:

* specific contraindication to statin therapy because of a previous coronary event or serum LDL-cholesterol levels > 190 mg/dL despite a low cholesterol (<200 mg/day) diet and a saturated fatty acid in take less than 7% of total calories will not be included
* chronic treatment with corticosteroids, nonsteroidal anti-inflammatory drugs, or immunosuppressive drugs
* acute myocardial infarction or cerebrovascular accident in the six months preceding the study - severe uncontrolled hypertension (diastolic blood pressure >115 and/or systolic blood pressure >220 mmHg)
* evidence or suspicion of renovascular disease, obstructive uropathy, type 1 diabetes mellitus, vasculitides, cancer
* elevated serum aminotransferase concentrations - chronic cough
* history of poor tolerance or allergy to ACEi, ATA or statins
* drug or alcohol abuse
* pregnancy, breast feeding and ineffective contraception
* legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the trial.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2003-03; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
24-hour urinary protein excretion rate, at the end of 6 months treatment phase | At 0, 2,3,4,5,6,7,8,9,10 months.

SECONDARY OUTCOMES:
Urinary protein/creatinine ratio; glomerular filtration rate (GFR); lipid profile. In a subgroup: renal plasma flow (RPF); filtration fraction albumin; IgG and IgM fractional clearance; insulin sensitivity; urinary endothelin excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Principal Investigator — Mario Negri Institute
Locations (16):
- Italy (16):
  - Hospital "Santa Maria della Gruccia" - Unit of Nephrology and Dialysis, Montevarchi, Arezzo
  - Clinical Research Center for Rare Diseases, Ranica, Bergamo
  - Hospital "S.Marte e S.Venere" - Unit of Nephrology and Dialysis, Acireale, Catania
  - Hospital "Vittorio Emanuele II, S. Bambino, Ferrarotto" - Unit of Nephrology and Dialisys, Catania, Catania
  - Hospital "Ciaccio" - Unit of Nephrolofy and Dialysis, Catanzaro, Catanzaro
  - Hospital "Santa Maria dell'Annunziata" - Unit of Nephrology, Bagno a Ripoli, Firenze
  - Hospital "Careggi Monna Tessa" - Unit of Nephrology and Dialysis, Florence, Firenze
  - Hospital "Casa Sollievo della Sofferenza" - Unit of Nephrology and Dialysis, San Giovanni Rotondo, Foggia
  - Hospital of Padova - Unit of Nephrology and Dialysis, Padua, Padova
  - Hospital "Civico e Benefratelli" - Unit of Nephrology and Hemodialysis, Palermo, Palermo
  - Hospital of Parma - Department of Medical Clinic, Parma, Parma
  - University of Sassari - Institute of Medical Pathology, Sassari, Sassari
  - Hospital "G.Mazzini" - Unit of Nephrology and Dialysis, Teramo, Teramo
  - Hospital "S.Giacomo Apostolo", Castelfranco Veneto, Treviso
  - Hospital of Mestre - Unit of Nephrology and Dialysis, Venezia, Venezia
  - "Ospedali Riuniti" CNR I.B.I.M. - Unit of Nephrology, Reggio Calabria

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Ruggenenti P, Perna A, Tonelli M, Loriga G, Motterlini N, Rubis N, Ledda F, Rota S Jr, Satta A, Granata A, Battaglia G, Cambareri F, David S, Gaspari F, Stucchi N, Carminati S, Ene-Iordache B, Cravedi P, Remuzzi G; ESPLANADE Study Group. Effects of add-on fluvastatin therapy in patients with chronic proteinuric nephropathy on dual renin-angiotensin system blockade: the ESPLANADE trial. Clin J Am Soc Nephrol. 2010 Nov;5(11):1928-38. doi: 10.2215/CJN.03380410. Epub 2010 Jul 29. PMID 20671225